CLINICAL TRIAL: NCT04437355
Title: Clinical, Functional and Radiological Outcome After Osteosynthesis of Ankle Fractures Using a Specific Provocation Test- a Combined Retro- and Prospective Study
Brief Title: Operative Treatment of Ankle Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spital Limmattal Schlieren (Other)
Responsible Party: Principal Investigator, Prof Urs Zingg, Head of Department of surgery, Spital Limmattal Schlieren
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-01124
Record Dates: First submitted 2020-01-07; First posted 2020-06-18 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Ankle Fracture, Trimalleolar; Ankle Fracture - Lateral Malleolus; Ankle Fracture, Bimalleolar
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Young and healthy Group of People (18-50 years) without any pathology of the lower limb
  Interventions: Diagnostic Test: Specific provocation test
- Ankle Fracture Type Weber B (Active Comparator): Young and healthy patients with an operative treated fracture of the ankle (type Weber B)
  Interventions: Diagnostic Test: Specific provocation test
- Ankle Fracture Weber C and complex (Active Comparator): Young and healthy patients with an operative treated fracture of the ankle (type Weber C or complex fracture)
  Interventions: Diagnostic Test: Specific provocation test

INTERVENTIONS:
Diagnostic Test: Specific provocation test — To compare the results the investigators invite a healthy control group matching in age and gender with the intervention cohort. The control group is informed about the study and asked to participate in the outpatient clinic. In case of informed consent, the participants are invited to the study site. The participants undergo the same provocation test of the ankle, and are asked to complete the specific provocation test. In case of substantial underachievement in the provocation test (<60% of maximum) an X-Ray of both ankles in a.p. and lateral projection is performed. The aim is to radiologically analyse the ankles, and to rule out any morphological reasons for the above mentioned underperformance.

SUMMARY:
Patients who underwent operative treatment of an ankle fracture with or without following removal of the osteosynthetic material are examined by a specific ankle provocation test, a questionnaire and X-Rays to evaluate the clinical, functional and radiological outcome compared to a healthy control group

DETAILED DESCRIPTION:
The study includes all patients operated from 09.12.2012 to 31.12.2020. Patients will undergo an X-Ray at least two years after primary surgery or at least one year after removal of the osteosynthetic material. The patients operated from 09.12.2012 to date are therefore a retrospective cohort, the patients from to date until 31.12.2020 a prospective cohort. This method is used to achieve the highest possible number of patients in a define period of time with no alteration of surgical technique.

All patients in the retrospective cohort are contacted at least 2 years after surgery (or 1 year after removal) via phone call or letter, informed about the study and asked to participate. In case of informed consent, they are invited to the study site. They are asked to complete the questionnaires and they undergo X-Ray of the affected and the non-affected ankle.

All patients in the prospective cohort are informed about the study and asked to participate in the outpatient clinic. In case of informed consent, they are invited to the study site at least 2 years after surgery. They are asked to complete the questionnaires and they undergo na X-Ray of the affected and non-affected ankle.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 and younger than 51 years
* Operative treatment of an ankle fracture
* Time operation to follow up: at least 2 years
* Time removal of osteosynthetic material to follow up: at least 1 year
* Time operative treatment to removal of the osteosynthetic material: at least 9 months
* Informed Consent as documented by signature (Appendix: Informed Consent Form)

Exclusion Criteria:

* Other pathologies of the lower limb of the affected and/or non-affected side (fractures, pre-existing arthrosis or operative treatment of the affected and/or non-affected limb)
* Pre-existing vascular (peripheral arterial disease, diabetes) or neurological diseases of the lower extremities
* Women who are pregnant
* Prevalence of an infection of the implanted osteosynthetic material

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Functional outcome | at least two year after surgery or one year after removal of the osteosynthetic material
  This outcome will be compared with a group of adults matching in terms of gender and age. Measured by:
  - a specific ankle provocation test: Multiple sport test measuring possible movement of the ankle and tolerating stress simulating in sportive movement such as weight bearing, leg press tests etc.
  The specific provocation test does not have a specific name, because it is self made.
Functional outcome | 24 months after initial operation
  This outcome will be compared with a group of adults matching in terms of gender and age. Measured by:
  - three questionnaires (quality of life, possible movement, restrictions in daily life etc.)

SECONDARY OUTCOMES:
Clinical outcome 1 | 24 months after initial operation
  - VAS: Visual analogue score 1-10
  Explanation: 1 means almost no pain, 10 is the worst pain one can imagine
Clinical outcome 2 | 24 months after initial operation
  - Quality of life questionnaire
  Explanation: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software for the commercial version, but no special software is needed for the RAND-36 version. Pricing depends on the number of scores that the researcher needs to calculate.
Clinical outcome 3 | 24 months after initial operation
  * Arthrosis compared to the non-affected ankle measured by X-Ray (after an ankle fracture followed by an operative Treatment)
  * The measurement consists of evaluation the joint congruency, quality of the bone and the cartilage and the clear spaces (medial, central, lateral).

OTHER OUTCOMES:
Specific ankle provocation test | 24 months after initial operation
  specific provocation test in our department of physiotherapy supervised by a physiotherapist and one of the investigators. measure of weight bearing, jump on one feet, balance.

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, Study Chair — Spital Limmattal Schlieren
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No